CLINICAL TRIAL: NCT05437263
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Oral Brepocitinib in Adults With Dermatomyositis
Brief Title: A Study to Investigate the Efficacy and Safety of Brepocitinib in Adults With Dermatomyositis
Acronym: VALOR
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Priovant Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PVT-2201-301; 2022-500367-12-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Dermatomyositis
Keywords: brepocitinib; dermatomyositis; TYK2/JAK1 inhibitor; PF-06700841; PVT-2201
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Brepocitinib Dose Level 1 PO QD (Experimental)
  Interventions: Drug: Brepocitinib
- Brepocitinib Dose Level 2 PO QD (Experimental)
  Interventions: Drug: Brepocitinib
- Placebo PO QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brepocitinib — Oral Brepocitinib
  Arms: Brepocitinib Dose Level 1 PO QD; Brepocitinib Dose Level 2 PO QD
Drug: Placebo — Oral Placebo
  Arms: Placebo PO QD

SUMMARY:
This is a phase 3, multicenter, randomized, placebo-controlled, double-blind study of treatment with brepocitinib (TYK2/JAK1 inhibitor) in adults with dermatomyositis (DM). The primary objective of this study is to assess the efficacy of two dose levels of brepocitinib in comparison to placebo, as measured by differences in the Total Improvement Score (TIS). After 52 weeks of double-blind treatment, participants have the option to continue therapy in a 52 week open-label extension phase where all participants will receive brepocitinib.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of dermatomyositis according to 2017 EULAR/ACR Classification Criteria for Idiopathic Inflammatory Myopathies
* Adult subjects (18-75 years old)
* Active muscle and skin disease at screening and baseline
* Prior therapy OR current therapy with corticosteroids, hydroxychloroquine, and/or one non-steroid immunosuppressant
* Weight > 40 kg to < 130 kg, and with a body mass index (BMI) < 40 kg/m2.

Exclusion Criteria:

* Dermatomyositis with end-stage organ involvement
* Dermatomyositis with irreversible muscle involvement
* History of:

  * Any lymphoproliferative disorder
  * Active malignancy;
  * History of cancer within 5 years prior to randomization (exceptions for basal cell carcinoma, squamous cell carcinoma, ductal carcinoma in situ of the breast, carcinoma in situ of the uterine cervix, or thyroid carcinoma.)
  * Cancer-associated dermatomyositis
* Overlap myositis/connective tissue disease (except for overlap with Sjögren's syndrome)
* Participants at a risk of thrombosis or cardiovascular disease
* Participants with a high risk for herpes zoster reactivation
* Participants with active or recent infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Total Improvement Score (TIS) at Week 52 | 52 weeks
  TIS is a composite endpoint based on improvement in the 6 Disease Activity Core Set Measure (CSM) scores and ranges from 0 to 100 (2016 American College of Rheumatology [ACR] Myositis Response Criteria/European League Against Rheumatism [EULAR]) where a higher score indicates more improvement

SECONDARY OUTCOMES:
Change from baseline in Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) Activity Score at Week 52 | 52 weeks
  CDASI Activity Score 0 to 100 with higher scores indicating a worse outcome.
Dermatomyositis Outcomes for Muscle and Skin (DMOMS) at Week 52 | 52 weeks
  DMOMS is a composite endpoint based on 4 component measures and ranges from 0 to 100 (Pandya, 2024) where a higher score indicates more improvement.
The proportion of participants achieving TIS ≥ 40 points (moderate improvement) at Week 52 | 52 weeks
Time to achievement of consecutive (≥ 2 visits) TIS ≥ 40 points (moderate improvement) by Week 52 | 52 weeks
The proportion of participants, regardless of baseline corticosteroid use, achieving TIS ≥ 40 points (moderate improvement) at Week 52 with 0 to ≤ 2.5 mg/day of oral prednisone (or equivalent) at both Week 48 and Week 52 | 52 weeks
The proportion of participants achieving ≥ 40% improvement with a ≥ 4-point improvement from baseline in CDASI Activity Score at Week 52 | 52 weeks
The proportion of participants achieving TIS ≥ 60 points (major improvement) at Week 52 | 52 weeks
Change from baseline in HAQ Disability Index score at Week 52 | 52 weeks
  Change from baseline in HAQ Disability Index score at Week 52. Health Assessment Questionnaire (HAQ) Disability Index: Score for function and disability from 0 [without any difficulty] to 3 [unable to do]. Higher score associated with worse outcome.
Change from baseline in CDASI Activity Score at Week 4 | 4 weeks

CONTACTS AND LOCATIONS:
Locations (101):
- United States (36):
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Scottsdale, Arizona
  - Clinical Trial Site, Irvine, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Denver, Colorado
  - Clinical Trial Site, Boynton Beach, Florida
  - Clinical Trial Site, Gainesville, Florida
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Plantation, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Augusta, Georgia
  - Clinical Trial Site, Marietta, Georgia
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Iowa City, Iowa
  - Clinical Trial Site, Kansas City, Kansas
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Ann Arbor, Michigan
  - Clinical Trial Site, Minneapolis, Minnesota
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, Manhasset, New York
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Oklahoma City, Oklahoma
  - Clinical Trial Site, Portland, Oregon
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Jackson, Tennessee
  - Clinical Trial Site, Austin, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Irving, Texas
- Argentina (3):
  - Clinical Trial Site, Quilmes, Buenos Aires
  - Clinical Trial Site, Caba, Buenos Aires F.D.
  - Clinical Trial Site, Mendoza
- Clinical Trial Site, Leuven, Belgium
- Bulgaria (2):
  - Clinical Trial Site, Plovdiv
  - Clinical Trial Site, Sofia
- Canada (2):
  - Clinical Trial Site, Vancouver, British Colombia
  - Clinical Trial Site, Newmarket, Ontario
- Chile (4):
  - Clinical Trial Site, Concepción, Región del Biobío
  - Clinical Trial Site, Recoleta
  - Clinical Trial Site, Santiago
  - Clinical Trial Site, Temuco
- Clinical Trial Site, Prague, Czechia
- Germany (5):
  - Clinical Trial Site, Mainz, Rhineland-Palatinate
  - Clinical Trial Site, Berlin
  - Clinical Trial Site, Dresden
  - Clinical Trial Site, Essen
  - Clinical Trial Site, Freiburg im Breisgau
- Hungary (3):
  - Clinical Trial Site, Debrecen
  - Clinical Trial Site, Pécs
  - Clinical Trial Site, Szeged
- Israel (5):
  - Clinical Trial Site, Ashkelon
  - Clinical Trial Site, Haifa
  - Clinical Trial Site, Poria – Neve Oved
  - Clinical Trial Site, Tel Aviv
  - Clinical Trial Site, Tel Litwinsky
- Italy (4):
  - Clinical Trial Site, Bari
  - Clinical Trial Site, Pavia
  - Clinical Trial Site, Roma
  - Clinical Trial Site, Torino
- Mexico (5):
  - Clinical Trial Site, Monterrey, Nuevo León
  - Clinical Trial Site, Mérida, Yucatán
  - Clinical Trial Site, Guadalajara
  - Clinical Trial Site, Mexico City
  - Clinical Trial Site, San Luis Potosí City
- Netherlands (2):
  - Clinical Trial Site, Nijmegen, Gelderland
  - Clinical Trial Site, Amsterdam
- Poland (6):
  - Clinical Trial Site, Bialystok, Podlaskie Voivodeship
  - Clinical Trial Site, Krakow
  - Clinical Trial Site, Lublin
  - Clinical Trial Site, Nowa Sól
  - Clinical Trial Site, Poznan
  - Clinical Trial Site, Warsaw
- Portugal (4):
  - Clinical Trial Site, Vila Nova de Gaia, Porto District
  - Clinical Trial Site, Guimarães
  - Clinical Trial Site, Lisbon
  - Clinical Trial Site, Porto
- Romania (2):
  - Clinical Trial Site, Bucharest
  - Clinical Trial Site, Cluj-Napoca
- Clinical Trial Site, Belgrade, Serbia
- South Korea (2):
  - Clinical Trial Site, Seoul
  - Clinical Trial Site, Suwon
- Clinical Trial Site, Madrid, Spain
- Taiwan (4):
  - Clinical Trial Site, Kaohsiung City
  - Clinical Trial Site, Taichung
  - Clinical Trial Site, Tainan
  - Clinical Trial Site, Taipei
- Turkey (Türkiye) (5):
  - Clinical Trial Site, Ankara
  - Clinical Trial Site, Antalya
  - Clinical Trial Site, Istanbul
  - Clinical Trial Site, Izmir
  - Clinical Trial Site, İzmit
- United Kingdom (3):
  - Clinical Trial Site, Bath
  - Clinical Trial Site, Manchester
  - Clinical Trial Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Priovant Therapeutics will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) from eligible studies upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Data requests will be reviewed and approved on the basis of scientific merit.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be made available within 24 months after study completion and will be accessible for a time frame appropriate for the approved proposal.
Access Criteria: Access will be provided following review and approval of a research proposal and execution of a Data Sharing Agreement (DSA). Further details on Priovant Therapeutics' data sharing criteria and process for requesting access can be obtained by emailing info@priovanttx.com.

REFERENCES:
- See also: Study Website — http://www.valorstudy.com